CLINICAL TRIAL: NCT07176078
Title: Evaluating the Added Benefit of Osteopathic Care to a Flexi-FODMAP Diet in Fibromyalgia Patients With Irritable Bowel Syndrome: a Randomized Sham-controlled Trial
Acronym: POISE-IBS-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25153_POISE-IBS-RCT
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Irritable Bowel Syndrome (IBS); Fibromyalgia (FM)
Keywords: Osteopathic Care; Irritable Bowel Syndrome; Fibromyalgia; FODMAP Diet
MeSH Terms: conditions — Irritable Bowel Syndrome; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic care + flexi FODMAP diet (Experimental)
  Interventions: Other: Osteopathic care; Behavioral: Flexi-FODMAP Diet
- Sham osteopathic care + flexi FODMAP diet (Sham Comparator)
  Interventions: Other: Sham Osteopathic care; Behavioral: Flexi-FODMAP Diet

INTERVENTIONS:
Other: Osteopathic care — Participants allocated to the osteopathic care group will receive 4 weekly consultations of person-centered osteopathic care. Each consultation will last approximately 45 minutes and consist of a careful medical history, a clinical examination, treatment, and advice (e.g. exercise, dietary, lifestyle).
  The osteopathic treatment protocol could be labeled as 'custom tailored': the determination of the treatment was left to the clinical judgment of the osteopath, meaning that no predefined, standardized osteopathic protocol would be implemented. Standard osteopathic techniques (Glossary of Osteopathic Terminology) can be applied, including diagnostic techniques (e.g. observation, neurological tests, palpation, and motion testing) and therapeutic direct (e.g. high-velocity low-amplitude, muscle energy), indirect techniques (e.g. strain counter strain, balanced ligamentous tension, balanced membranous tension), or combined techniques.
  Arms: Osteopathic care + flexi FODMAP diet
Other: Sham Osteopathic care — For this trial, sham intervention will mimic the osteopathic care according to the "touch equality assumption". Therefore, it mimics a clinical examination and treatment. The sham clinical evaluation involves a full evaluation of the position and mobility of the spine.This screening of the patient will be performed using conventional osteopathic manual tests, without any intention to make a diagnosis. Sham treatment will involve light manual contact, with the subject lying supine on the treatment table.
  Arms: Sham osteopathic care + flexi FODMAP diet
Behavioral: Flexi-FODMAP Diet — In addition to the real or sham osteopathic care, all participants will follow a 4-week flexi-FODMAP diet delivered online. Participants will receive structured dietary instructions via a customized online platform, based on the NHS Gentle-FODMAP diet guidelines and informed by expert input from dieticians. This modified "FODMAP-gentle" approach involves a targeted, less restrictive elimination of selected high-FODMAP foods.

SUMMARY:
Dietary modifications are often recommended as first-line treatment for irritable bowel syndrome, with the FODMAP diet being the most effective intervention to improve global gastrointestinal symptoms. Due to the heterogeneity of symptoms, patients often seek complementary or alternative therapies. This randomized clinical trial aims to determine whether osteopathic care provides additional improvement in gastrointestinal symptoms compared to sham osteopathic care, when both are combined with a flexible FODMAP diet. The trial will also assess the safety and tolerability of osteopathic care.

The main questions it aims to answer are:

Does osteopathic care reduce IBS symptom severity more than sham osteopathic care?

Does osteopathic care improve pain, quality of life, anxiety, fatigue, work productivity, and gut microbiota compared to sham osteopathic care?

Do participants adhere to the flexible FODMAP diet and osteopathic care, and are the effects of osteopathic care maintained at 3- and 6-months post-intervention?

Can pretreatment factors, such as sociodemographic characteristics, IBS severity, predominant symptoms, psychological state, or gut microbiota composition, predict response to osteopathic care?

What adverse effects occur with osteopathic care compared to sham care?

Participants will:

Visit the osteopathy clinic to receive four sessions of real or sham osteopathic care

Complete online assessments before and after the intervention, and at 3- and 6-months post-intervention

Provide stool samples before and after the four osteopathic or sham sessions

Keep a three-day food diary and a ten-day stool diary before and after the intervention, and at 3- and 6-months post-intervention

ELIGIBILITY:
Inclusion Criteria:

This study includes participants who meet the following criteria:

1. are over 18 years old;
2. have a diagnosis of IBS by a medical doctor according to the Rome IV criteria and have an IBS-SSS score of ≥175 (indicating moderate to severe IBS symptoms);
3. have a medical diagnosis of fibromyalgia or meet the 2016 American College of Rheumatology criteria, characterized by chronic (≥3 months) widespread pain(i.e., a Widespread Pain Index(WPI) score of ≥7 with a Symptom Severity Score of ≥5, or a WPI score of 4-6 with a Symptom Severity Score ≥9 on the Widespread Pain Index).

Participants will be allowed to use probiotic products and follow a lactose-reduced diet, as long as they kept their usual intake throughout the study, unless a further reduction in lactose was recommended for those assigned to diet therapy. IBS medications, including antidepressants, will be allowed if used consistently at a stable dose for at least 2-3month prior to inclusion. Additionally, participants will need to be willing to adjust their current dietary habits in order to take part in the study.

Exclusion Criteria:

This study excludes participants who meet any of the following criteria:

1. have other gastrointestinal disorders (e.g., inflammatory bowel disease, celiac disease) that could explain the current symptoms;
2. have diseases affecting gastrointestinal function, including a history of bariatric surgery;
3. have allergies or food hypersensitivity (other than lactose intolerance);
4. have any major dietary restrictions or food allergies;
5. are pregnant or planning pregnancy during the trial (within the next seven months);
6. have a BMI ≤18 kg/m²; or 7) have received osteopathic care for IBS and/or are already following the FODMAP dietary intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) | Baseline and after 4 weeks (post-intervention)
  The IBS Symptom Severity Score (IBS-SSS) will be utilized to evaluate the severity of IBS symptoms. This scale provides an overall score ranging from 0 to 500, with higher scores indicating greater symptom severity. The questionnaire includes the following components: intensity and frequency of abdominal pain, abdominal distension, dissatisfaction with bowel habits, and the overall impact of IBS on daily life ("life interference"). Scores are categorized as follows: 75-175 indicates mild severity, 175-300 represents moderate severity, and 300 or above reflects severe symptoms. The IBS-SSS considered a valid and reliable scale, with a Cronbach's Alpha = 0.80.

SECONDARY OUTCOMES:
Change in Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The IBS Symptom Severity Score (IBS-SSS) will be utilized to evaluate the severity of IBS symptoms. This scale provides an overall score ranging from 0 to 500, with higher scores indicating greater symptom severity. The questionnaire includes the following components: intensity and frequency of abdominal pain, abdominal distension, dissatisfaction with bowel habits, and the overall impact of IBS on daily life ("life interference"). Scores are categorized as follows: 75-175 indicates mild severity, 175-300 represents moderate severity, and 300 or above reflects severe symptoms. The IBS-SSS considered a valid and reliable scale, with a Cronbach's Alpha = 0.80.
3 day dietary dairy | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The diary asks for dietary intake information of two weekdays and one day in the weekend. Collected data with the 3-day food diary will allow us to find out approximate calorie intake, micronutrient intake, macronutrient intake of each participant.
Stool Diary | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The patients will record all bowel movements over a 10-day period using a stool diary, based on the Bristol Stool Form (BSF) scale. The diary will document stool frequency (number of stools per day), mean stool consistency on a 7-point scale, and will be used to classify IBS subtypes and evaluate bowel habits. Sub-types of IBS are divided into four categories based on the predominant stool form; IBS with predominant constipation (IBS-C, ≥25% hard stools (BSF 1 or 2) and <25% loose stools (BSF 6 or 7)), IBS with predominant diarrhea (IBS-D, ≥25% loose stools and <25% hard stools), IBS with alteration between constipation and diarrhea (IBS-M, ≥25% of reported stools hard and ≥25% loose); and un-subtyped IBS (IBS-U, insufficient abnormality of stool consistency to meet criteria for IBS-C, -D, or -M).
Change in Pain intensity | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The "Brief Pain Inventory" allows to rate the worst pain in the last 24 hours, the least pain in the last 24 hours, the average pain and the pain intensity at the moment of filling out the questionnaire. This tool also assesses the interference of pain with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep via an 11-point numeric rating pain scale, ranging from 0 (no pain) to 10 (worst pain)
Change in Fatigue severity | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The Multidimensional Fatigue Inventory-20 (MFI-20) assesses the severity of general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue. Each dimension contains 4 questions, with a range of scores between 4 and 20, generating a total score between 0 and 100. A higher score indicates more severe fatigue. The MFI-20 is considered a valid and reliable scale, with a Cronbach's Alpha = 0.93.
Change in Irritable Bowel Syndrome related quality of Life | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The IBS quality of Life (IBS-QoL) is an IBS-specific QoL questionnaire that measures 10 domains that have been found to be relevant to patients with IBS: emotional health, mental health, health belief, sleep, energy, physical functioning, diet, social role, physical role, and sexual relations. The minimum score is 30 and the maximum score is 160. The higher the score, the better the QoL. The IBS-QoL is considered a valid and reliable scale, with Cronbach alpha=0.95.
Change in Gastrointestinal-Specific symptom anxiety | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The Visceral Sensitivity Index measures GI-specific anxiety, that is, anxiety originating from fear of GI symptoms, which is related to the unpredictable symptom pattern commonly found in IBS. Each item can be scored from one, 'strongly agree', to six, 'strongly disagree'. High-sum scores represent more severe GI-specific anxiety. The Visceral Sensitivity Index is considered a valid and reliable scale, with a Cronbach's Alpha = 0.92.
Change in Depression | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The Patient Health Questionnaire (PHQ-9) will be used to diagnose depressive disorders. The PHQ-9 measures the severity of a depressive disorder with nine questions resulting in a sum score between 0 and 27 points. A score of 5 or more indicates mild depression, from 10 moderate, from 15 moderate-severe and above 20 severe depression. The internal and test-retest reliabilities of the PHQ-9 were both excellent, with a Cronbach's α of 0.89.
Change in Sleep Quality | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  Sleep quality experienced in the previous month were measured using the 19-item self-reported Pittsburgh Sleep Quality Index (PSQI). The 19-items generate seven component scores: subjective sleep quality, sleep latency, sleep duration (i.e., quantity), habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each of these seven component scores is weighted equally on a scale ranging from 0 to 3, 0 indicating no difficulty and 3 indicating severe difficulty. Overall, sleep quality (global PSQI score) was calculated by summing the seven component scores, which range from 0 (better) to 21 (worse); a global PSQI score > 5 is consistent with poor sleep quality. The internal and test-retest reliabilities of the PSQI were both excellent, with a Cronbach's α of 0.83.
Change in Perceived stress | Baseline and after 4 weeks (post-intervention)
  Perceived stress was measured using the PSS, which also measured participants' current stress levels and which situations in their lives were appraised as stressful. The PSS is a 10-item questionnaire where individuals are asked about their feelings in the past month; it is scored on a 5-point scale ranging from 0 (Never) to 4 (Very often). Four PSS responses are then reverse-scored, and a sum is calculated to obtain a total, where higher scores suggest higher perceived stress. The scale validity is strong (r = 0.72), as is the test-retest reliability (r = 0.93, p < 0.001).
Change in Work Productivity and Activity | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  The Work Productivity and Activity Impairment Questionnaire-IBS measures whether IBS symptoms affect the ability to work and perform everyday activities with four different variables: absenteeism, presenteeism, overall work impairment, and activity impairment. Each variable ranges from 0% to 100%, with higher values indicating higher impairment. The Work Productivity and Activity Impairment Questionnaire-IBS is a valid and reliable scale with high test-retest correlations (r = 0.97 - 0.99).
Change in microbiota content | Baseline and after 4 weeks (post-intervention)
  Fecal microbiota analysis
Adherence to allocated intervention | Baseline, after 4 weeks (post-intervention), 3 months after the end of intervention, and 6 months after the end of intervention
  Dietary intervention (4 weeks): Adherence assessed through participant-completed food diaries and questionnaire. Patients will rate the number of times they forgot to follow the diet on a Likert scale (0 = never to 6 = constantly)
  Osteopathy care (4 weeks): Adherence monitored using attendance records of scheduled sessions.
  Long-term follow-up: Adherence evaluated through patient diaries focusing on maintenance of dietary recommendations and osteopathy-related practices.
Patient Satisfaction | After 4 weeks (post-intervention)
  Treatment satisfaction was scored as an improvement in IBS symptoms compared with baseline and ranging from 'a lot worse' (zero) to 'extremely better' (seven).
  Additionally, patient attending the osteopathic care, the level of satisfaction will be assessed at the end of the study by asking patients their global appreciation of osteopathic care and whether they would agree to pay for subsequent manipulative procedures.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancini JD, Yao S, Martinez LR, Shakil H, Li TS. Gut Microbiome Changes with Osteopathic Treatment of Constipation in Parkinson's Disease: A Pilot Study. Neurology (ECronicon). 2021 Feb;13(2):19-33. Epub 2021 Jan 30. PMID 33899052
- [Background] Buffone F, Tarantino AG, Belloni F, Spadafora A, Bolzoni G, Bruini I, Bergna A, Vismara L. Effectiveness of Osteopathic Manipulative Treatment in Adults with Irritable Bowel Syndrome: A Systematic Review and Meta-Analysis. Healthcare (Basel). 2023 Aug 31;11(17):2442. doi: 10.3390/healthcare11172442. PMID 37685480
- [Background] Attali TV, Bouchoucha M, Benamouzig R. Treatment of refractory irritable bowel syndrome with visceral osteopathy: short-term and long-term results of a randomized trial. J Dig Dis. 2013 Dec;14(12):654-61. doi: 10.1111/1751-2980.12098. PMID 23981319
- [Background] Florance BM, Frin G, Dainese R, Nebot-Vivinus MH, Marine Barjoan E, Marjoux S, Laurens JP, Payrouse JL, Hebuterne X, Piche T. Osteopathy improves the severity of irritable bowel syndrome: a pilot randomized sham-controlled study. Eur J Gastroenterol Hepatol. 2012 Aug;24(8):944-9. doi: 10.1097/MEG.0b013e3283543eb7. PMID 22546751